CLINICAL TRIAL: NCT03091569
Title: Effects of VITAmin K in Lessening Erythema Grade Associated to Injection Site Reactions in Patients Treated With PlegridY (VITALITY)
Brief Title: Effects of Vitamin K on Redness Associated With Injection Site Reactions in Participants Treated With Plegridy
Acronym: VITALITY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: ITA-PEG-15-10859
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin K (Active Comparator)
  Interventions: Other: Vitamin K Cream
- Control (Placebo Comparator)
  Interventions: Other: Placebo Cream

INTERVENTIONS:
Other: Vitamin K Cream — To be applied topically 3 times in 24 hours (approximately at 8 and 16 hours post initial application) from the appearance of the erythema.
  Other Names: Filloskin K1
  Arms: Vitamin K
Other: Placebo Cream — To be applied topically 3 times in 24 hours (approximately at 8 and 16 hours post initial application) from the appearance of the erythema.
  Arms: Control

SUMMARY:
The primary objective of the study is to investigate whether topical Vitamin K application reduces the grade of erythema in comparison with a vehicle cream (placebo) through physicians' assessment and participant self-assessment.

The secondary objectives of this study are to evaluate in this study population: effects of Vitamin K in reducing the burning sensation and local pain; effects of Vitamin K in reducing the erythema diameter; and the evaluation of participants' satisfaction related to the injection treatment.

ELIGIBILITY:
Key Inclusion Criteria:

* Relapsing-Remitting Multiple Sclerosis (RRMS) participants for which Plegridy is deemed necessary by the neurologist. Participants switching from other Disease Modifying Treatments (DMTs) will be eligible provided that Plegridy is administered at an injection site different from the previous one.

Key Exclusion Criteria:

* Participants with other skin disorders
* Pregnancy or current breast-feeding
* Depression and other psychiatric disorders
* Unwillingness or inability to comply with the requirements of the protocol.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-03-10 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Change in Clinician's Erythema Assessment (CEA) scale from pre-application of topical cream to 24 hours post-application | Week 4, week 6, and week 8
  Erythema (redness) evaluated at the site of injection by the clinician on a scale of 0 (clear) to 4 (severe)
Change in Participants Erythema Self-Assessment (PSA) scale from pre-application of topical cream to 24 hours post-application | Week 4, week 6, and week 8
  Erythema (redness) at the site of injection rated by the participant on a scale of 0 (clear) to 4 (severe)

SECONDARY OUTCOMES:
Change in Visual Analogue Scale (VAS) score from pre-application of topical cream to 24 hours post-application | Week 4, week 6, and week 8
  Severity of local pain and burning assessed by the participant on a scale of 0 (no discomfort) to 10 (maximum discomfort imaginable)
Change in Adapted Multiple Sclerosis Treatment Concerns Questionnaire (MSTCQ) from pre-application of topical cream to 24 hours post-application | Week 4, week 6, and week 8
  Adapted MSTQC self-administered questionnaire evaluates the sum of scores for the "injection systems satisfaction" section questions 1-9 and the "side effects" section questions 1-11, with a minimum possible total score of 20 and a maximum possible total score of 100. Lower total scores indicate better outcomes.
Change in the longest diameter of erythema from pre-application of topical cream to 24 hours post-application | Week 4, week 6, and week 8
  Measured by the physician using a ruler before and 24 hours after the topical application of cream

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Napoli, Italy